CLINICAL TRIAL: NCT00979004
Title: A Phase 2, Multi-Center, Single-Blind, Placebo-Controlled Pharmacodynamic Evaluation of ICA-105665 in Epilepsy Patients With a Photo-Induced Paroxysmal EEG Response
Brief Title: A Study to Investigate the Effect of ICA-105665 in Photosensitive Epilepsy Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated on September 12, 2010 per protocol following a serious adverse event that occurred with the first subject dosed at 600 mg.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ICA-105665-04; B5311005
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-09

CONDITIONS: Epilepsy
Keywords: Photosensitivity; Epilepsy; Seizures
MeSH Terms: conditions — Epilepsy; Photosensitivity Disorders; Seizures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- ICA-105665 (Experimental)
  Interventions: Drug: ICA-105665

INTERVENTIONS:
Drug: ICA-105665 — Oral tablet. Dose forms of 50 and 100 mg or placebo will be used. A single dose will be administered that can range from placebo or 100 to 600 mg.

SUMMARY:
Subjects with epilepsy with a documented photoparoxysmal response to intermittent photic stimulation (IPS) will participate. Four subjects will be enrolled at each dose level and will receive a single dose of placebo and a single dose of ICA-105665 during the study, each followed by intermittent photic stimulation. The effects of ICA-105665 on the photoparoxysmal electroencephalography (EEG) response of each group will be reviewed before the dose is selected for each subsequent group of subjects.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis and history of epilepsy for which they are on 0-2 concurrent antiepileptic drugs.
* On a stable dose of their current AED(s) for 4 weeks prior to the Screening Visit.
* Must be in good health (with the exception of epilepsy), as determined by the Primary Investigator via the medical history, a physical examination, and screening laboratory investigations.
* A body mass index (BMI) between 18 and 35.
* Able and willing to give written informed consent prior to participation in the study.
* A reproducible IPS-induced photo-paroxysmal EEG response (PPR) of at least 3 points on a frequency assessment scale in at least one eye condition and no change of more than 3 frequencies in 2 repeated measurements recorded at the Screening Visit.

Exclusion Criteria:

* History of non-epileptic seizures (metabolic, structural, or pseudoseizures).
* History of status epilepticus while on any antiepileptic medication.
* The etiology of the seizures is due to any of the following; progressive degenerative disease, metabolic illness, active infection, demyelination, drugs, alcohol.
* The subject has used benzodiazepines (oral, intra-muscular, or suppository) as escape medication within the past 6 months.
* The subject has taken an investigational medication within 30 days prior to the Day 1.
* Women who are pregnant or lactating.
* An active Central Nervous System (CNS) infection, demyelinating disease, degenerative neurological disease or any CNS disease deemed to be progressive during the course of the study that may confound the interpretation of the study results.
* The subject has a clinically significant (e.g., cancerous, unstable, progressive, functionally disabling, or infectious) medical condition that would interfere with the ability to complete the study or that might interfere with the absorption, distribution, metabolism, and/or excretion of drugs.
* Subjects with impaired hepatic function [ALT (Alanine aminotransferase), AST (Aspartate aminotransferase) =3 times the upper limit of normal] or any clinically significant laboratory abnormality that, in the opinion of the investigator, would increase the risk of participation or interfere with the interpretatio of the study results.
* History of alcoholism, drug abuse, or drug addiction within the last 12 months.
* Clinically significant psychiatric illness, psychological or behavioral problem which, in the opinion of the investigator would interfere with the subject's ability to participate in the study OR the subject is receiving therapy with neuroleptic drugs.
* Subject experiences a clinical seizure during any IPS procedure performed during the screening period.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Change in photosensitivity response | begin 1 hr post dose for 8 hours

SECONDARY OUTCOMES:
To correlate plasma concentrations of ICA-105665 with effect on the frequency range of IPS-induced PPR (Photoparoxysmal response) in subjects with photosensitive epilepsy. | 3 days
To assess the safety of a single dose of ICA-105665 in subjects with photosensitive epilepsy. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Chesterfield, Missouri
  - Pfizer Investigational Site, Nashville, Tennessee

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=ICA-105665-04&StudyName=A%20Study%20to%20Investigate%20the%20Effect%20of%20ICA-105665%20in%20Photosensitive%20Epilepsy%20Patients